CLINICAL TRIAL: NCT06522308
Title: Prevalence of Cholelithiasis in Patients Presenting with Umbilical Hernia, and Vice Versa: Prospective Multicenter Cross-sectional Study
Brief Title: Prevalence of Cholelithiasis with Umbilical Hernia
Status: Completed | Type: Observational
Sponsor: Konya Meram State Hospital (Other)
Responsible Party: Principal Investigator, Alpaslan Şahin, Principal investigator, Konya Meram State Hospital
Other Study IDs: Hernia Study Group
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-10

CONDITIONS: Umbilical Hernia; Cholelithiasis
MeSH Terms: conditions — Hernia, Umbilical; Cholelithiasis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cholelithiasis Group: It is determined whether there is an umbilical hernias in patients with cholelithiasis
  Interventions: Diagnostic Test: Umbilical region superficial tissue ultrasound
- Umbilical Hernia Group: It is determined whether patients with umbilical hernia have cholelithiasis or not.
  Interventions: Diagnostic Test: Hepatobiliary ultrasound

INTERVENTIONS:
Diagnostic Test: Hepatobiliary ultrasound — The presence of cholelithiasis in patients with umbilical hernia is detected by hepatobiliary ultrasound
  Groups: Umbilical Hernia Group
Diagnostic Test: Umbilical region superficial tissue ultrasound — The presence of umbilical hernia in patients with cholelithiasis is detected by ultrasound of the superficial tissue of the umbilical region.
  Groups: Cholelithiasis Group

SUMMARY:
Researchers aim to determine the exact prevalence and risk factors for the association of gallstones and umbilical hernia. Umbilical hernia is defined according to the European Hernia Society Classification for primary and incisional abdominal wall hernias as hernias occurring from 3 cm above to 3 cm below the umbilicus. The main outcome measures are the presence of gallstones in patients presenting with umbilical hernia and the presence of umbilical hernia in patients diagnosed with gallstones. Patients with umbilical hernia are examined with biliary ultrasound, while patients with cholelithiasis are evaluated for umbilical hernia by physical examination and ultrasound. Factors such as age, gender, body mass index (BMI), family history, comorbidities, tobacco use, parity, and history of multiple pregnancy are analyzed as potential risk factors.

DETAILED DESCRIPTION:
Umbilical hernia and cholelithiasis are quite common in general surgical practice. The coexistence of cholelithiasis and umbilical hernia has been previously reported in the literature. However, most of the publications on this subject are retrospective series, and the prevalence of cholelithiasis in patients with umbilical hernia and the risk factors of umbilical hernia in patients with cholelithiasis have not been investigated prospectively to date. This study aims to fill this gap by providing prospective data on the prevalence and risk factors associated with the coexistence of these conditions.

Researchers aim to determine the exact prevalence and risk factors for the association of gallstones and umbilical hernia. Umbilical hernia is defined according to the European Hernia Society Classification for primary and incisional abdominal wall hernias as hernias occurring from 3 cm above to 3 cm below the umbilicus. The main outcome measures are the presence of gallstones in patients presenting with umbilical hernia and the presence of umbilical hernia in patients diagnosed with gallstones. Patients with umbilical hernia are examined with biliary ultrasound, while patients with cholelithiasis are evaluated for umbilical hernia by physical examination and ultrasound. Factors such as age, gender, body mass index (BMI), family history, comorbidities, tobacco use, parity, and history of multiple pregnancy are analyzed as potential risk factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with umbilical hernia
* Patients with cholelithiasis

Exclusion Criteria:

* Having previously had surgery for an umbilical hernia
* Having undergone abdominal surgery with a median line incision
* having collagen tissue disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All female and male cholelithiasis patients and umbilical hernia patients over the age of 18 who applied during the research period constitute the study population.
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Presence of cholelithiasis in umbilical hernia patients | 2 days
  In umbilical hernia patients, the presence of cholelithiasis is determined by hepatobiliary ultrasound.
Presence of umbilical hernia in cholelithiasis patients | 2 days
  In patients with cholelithiasis, the presence of umbilical hernias is determined by superficial tissue ultrasound of the umbilical region.

SECONDARY OUTCOMES:
Body mass index | 2 days
  Body mass index is calculated by dividing kilograms by height squared (kilograms / height squared).
The female-male ratio | 2 days
  The female-male ratio is found by the number of females divided by the number of males (female/male ratio).
Concomitant diseases ratio | 2 days
  It is found by dividing the number of patients with comorbidities by the total number of patients

CONTACTS AND LOCATIONS:
Overall Officials: Alpaslan Sahin, MD, Principal Investigator — Konya Meram State Hospital
Locations (1):
- Konya Training and Research Hospital, Konya, Turkey (Türkiye)